CLINICAL TRIAL: NCT02102750
Title: A Phase I Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Preservative Free Tafluprost Ophthalmic Solution (0.0015%) in Pediatric Patients Diagnosed With Glaucoma or Ocular Hypertension
Brief Title: A Study to Evaluate Pharmacokinetics of Tafluprost Ophthalmic Solution (0.0015%) in Pediatric Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santen Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201350; 2013-004302-26 (EudraCT Number)
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tafluprost (Experimental)
  Interventions: Drug: Preservative free tafluprost opthalmic solution

INTERVENTIONS:
Drug: Preservative free tafluprost opthalmic solution — 0.0015% eye drops q.d, in both eyes for 7 to 9 days

SUMMARY:
The purpose of the study is to examine how preservative free tafluprost ophthalmic solution (0.0015%) is distributed in blood circulation after ocular administration in children who have glaucoma or elevated intraocular pressure. Tolerance to the drug and safety in general will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a non-smoking male or female ≤ 17 years of age on the day of signing the informed consent. Infants must be at least 1 month of age
* A diagnosis of primary or secondary pediatric glaucoma or ocular hypertension in one or both eyes
* A history of IOP greater than or equal to 22 mmHg in at least one eye. Newly diagnosed patients may have this criterion fulfilled at the pre-study visit.
* Patient is currently prescribed ocular hypotensive medication and who according to investigator's judgement may discontinue the use at least day before the Day 1 visit, or patient is treatment-naïve (those who have never used used ocular hypotensive medication).
* Female patients of reproductive potential must demonstrate a negative pregnancy test at the pre-study visit
* Patient is judged to be in good health, other than having glaucoma or ocular hypertension, based on medical history, physical examination, vital signs measurements, and laboratory safety tests performed at the pre-study visit and/or prior to administration of the initial dose of study drug
* Patient has no clinically significant abnormality on electrocardiogram (ECG) performed at the pre-study visit
* Parent/legal guardian and/or patient have/has provided a written informed consent (according to existing local regulations) and patient assent has been given as applicable.
* The patient and parent/guardian should agree to comply with study restrictions, treatment plan, procedures and keep scheduled clinic visits.

Exclusion Criteria:

* Patient currently wears continuous wear contact lenses (use of daily wear contact lenses during the study is permitted)
* One-sighted or monocular patients, including patients who cannot be dosed in both eyes for any reason
* History of goniotomy or trabeculotomy within 1 month of pre-study visit or history of cataract surgery, laser surgery, filtration surgery, implant surgery or cyclodestructive surgery within 3 months prior to pre-study visit in one or both eyes.
* Patient has a history or evidence of significant ocular trauma within 3 months of prestudy visit
* Patient has a history or evidence of recent ocular inflammation and/or infection within 1 month of pre-study visit
* Patient has chronic conjunctivitis, chronic keratitis or lacrimal deficiency
* Patient is pregnant, breastfeeding, expecting to conceive within the projected duration of the study
* Patient has had major (non-ocular) surgery, loss of > 5 cc/kg of blood within 4 weeks of the pre-study visit
* Any other ocular, systemic or psychiatric disease/condition or laboratory abnormality
* History of febrile illness within 5 days prior to start of study treatment
* Patient has a history of hypersensitivity to any component of tafluprost eye drops, or known severe or serious hypersensitivity to any prostaglandin analogue product (e.g. latanoprost)
* Patient has a history of multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription (over-the-counter) drugs or food
* There is any concern by the investigator regarding the safe participation of a patient in the study
* Current participation in another clinical trial involving an investigational drug/device, or participation in such a trial within the last 30 days from the pre-study visit

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05-29 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of tafluprost acid. | 8 days +/- 1 day window

CONTACTS AND LOCATIONS:
Overall Officials: Auli Ropo, Study Director — Santen Oy
Locations (2):
- Childrens Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania, United States
- Moorfields Eye Hospital, London, United Kingdom